CLINICAL TRIAL: NCT04478708
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 133 in Subjects With Obesity
Brief Title: Single and Multiple Ascending Dose Study of AMG 133 in Participants With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20180048
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: maridebart cafraglutide (Experimental): Up to 7 single ascending dose cohorts (cohorts 1 to 6 and cohort 11).
  Interventions: Biological: maridebart cafraglutide
- Part A: Placebo (Placebo Comparator): Up to 7 single ascending dose cohorts (cohorts 1 to 6 and cohort 11).
  Interventions: Drug: Placebo
- Part B: maridebart cafraglutide (Experimental): Up to 4 multiple ascending dose cohorts (cohorts 7 to 10).
  Interventions: Biological: maridebart cafraglutide
- Part B: Placebo (Placebo Comparator): Up to 4 multiple ascending dose cohorts (cohorts 7 to 10).
  Interventions: Drug: Placebo
- Part C: maridebart cafraglutide (Experimental): Up to 2 open-label, multiple ascending dose cohorts (cohorts 12 to 13) treated with doses previously studied in Part A and Part B.
  Interventions: Biological: maridebart cafraglutide

INTERVENTIONS:
Biological: maridebart cafraglutide — Participants will receive maridebart cafraglutide as a single dose in Part A and multiple doses in Part B and C.
  Arms: Part A: maridebart cafraglutide; Part B: maridebart cafraglutide; Part C: maridebart cafraglutide
Drug: Placebo — Participants will receive placebo as a single dose in Part A and multiple doses in Part B.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The study aims to assess the safety and tolerability of maridebart cafraglutide as single and multiple doses in participants with obesity

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent before initiation of any study-specific activities/procedures.
* Age ≥ 18 years to ≤ 65 years, at the time of signing the informed consent.
* Except for obesity, otherwise healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and ECGs on day -2 (cohorts 1-6, cohort 11-13) or day -1 (cohorts 7-10) and screening.
* Body mass index between ≥ 30.0 kg/m^2 and ≤ 40.0 kg/m^2.
* Have a stable body weight (< 5 kg self-reported change during the previous 8 weeks) before screening.
* Willing to maintain current general diet and physical activity regimen, except for the physical activity in the 72 hours before each blood sample collection for the clinical laboratory analysis, which should not be strenuous.
* Females must be of nonreproductive potential

  • Postmenopausal as defined as:
* Age of ≥ 55 years with no menses for at least 12 months; OR
* Age < 55 years with no menses for at least 12 months AND with a follicle-stimulating hormone level > 40 IU/L or according to the definition of "postmenopausal range" for the laboratory involved; OR

  * History of hysterectomy; OR
  * History of bilateral oophorectomy.
* For patients in cohorts 7-10 only, participants must have a smartphone device with the capability of downloading apps or other digital tools required for this cohort.

Exclusion Criteria:

* History or clinical evidence of diabetes mellitus, including hemoglobin A1c (HbA1c) > 6.5% and/or a fasting glucose ≥ 125 mg/dl (6.9 mmol/L) at screening.
* Triglycerides ≥ 5.65 mmol/L (ie, 500 mg/dL) at screening.
* Screening calcitonin ≥ 50 ng/L.
* Hepatic liver enzymes aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, or total bilirubin levels > 1.5 times the upper limit of normal (ULN) at screening. If ALT is > 1.5 x the ULN at screening AND the AST, alkaline phosphatase, and total bilirubin levels are within normal limits, then participant may be eligible for enrollment after a discussion with the medical monitor.
* History or clinical evidence of bleeding diathesis or any coagulation disorder, including prothrombin time (PT), activated partial thromboplastin time (PTT), international normalized ratio (INR), or platelet count outside of the laboratory's normal reference range at screening. If a single value (PT, PTT, INR, or platelet count) is outside the normal reference range at screening and the participant does not have evidence of any other bleeding or coagulation disorder, then the participant may be eligible for enrollment after a discussion with the medical monitor.
* History of gastrointestinal abnormality that could affect gastrointestinal motility (including small bowel or colonic resection, inflammatory bowel disease, irritable bowel disease, and colon or gastrointestinal tract cancer).
* Participants with a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 or a personal history of nonfamilial medullary thyroid carcinoma.
* Participants with a history of confirmed chronic pancreatitis or idiopathic acute pancreatitis.
* Participants with a history of gall bladder disease (ie, cholelithiasis or cholecystitis) not treated with cholecystectomy.
* Untreated or uncontrolled hypothyroidism/hyperthyroidism defined as thyroid stimulating hormone > 6 mIU/L or <0.4 mIU/L.
* A corrected QT interval (QTc) at screening of > 450 msec in males or > 470 msec in females or history of long QT syndrome.
* Participants with a history of renal impairment or renal disease and/or estimated glomerular filtration rate ≤ 60 mL/min/1.73 m^2.
* Obesity induced by other endocrinologic disorders (eg, Cushing's Syndrome).
* Previous surgical treatment for obesity (excluding liposuction if performed >1 year before study entry) and/or participants with recent (within 6 months) or planned endoscopic treatment for obesity.
* History of major depressive disorder.
* History of other severe psychiatric disorders, eg schizophrenia, bipolar disorder.
* Any lifetime history of a suicidal attempt or of any suicidal behavior.
* Surgery scheduled for the study duration period, except for minor surgical procedures, at the discretion of the investigator.
* Positive results for human immunodeficiency virus antibodies, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C virus RNA. For hepatitis C, hepatitis C antibody testing is done at screening, followed by hepatitis C virus RNA by polymerase chain reaction if hepatitis C antibody is positive.
* Systolic blood pressure ≥ 150 mm Hg or diastolic blood pressure ≥ 90 mm Hg at screening, or on day -2. For each visit, if the initial blood pressure is elevated, the reading may be repeated once at least 15 minutes later and the lower of the 2 readings may be used.
* History of malignancy of any type, other than in situ cervical cancer or surgically excised nonmelanomatous skin cancers occurring more than 5 years before randomization.
* Use of the following agents are excluded unless there is a prior consultation between the investigator and Amgen medical monitor:

  * Prescription and nonprescription drugs within 14 days or 5 half-lives, whichever is longer, before the first dose of investigational product, with exception of hormone replacement therapy (eg, estrogen, thyroid).
  * All herbal medicines, vitamins, and supplements within 30 days before receiving the first dose of investigational product.
  * Exceptions must be reviewed and approved by the investigator and Amgen medical monitor. Written documentation of this review and Amgen acknowledgment is required for participant participation.
* Current or history of treatment with medications that may cause significant weight gain or loss, within 3 months before screening, including systemic corticosteroids (except for a short course of treatment, ie, 7 to 10 days), tricyclic antidepressants, atypical antipsychotic and mood stabilizers (eg, imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid and its derivatives, and lithium).
* Current participation (or within the last 3 months) in an organized weight reduction program or currently using or used within 3 months before screening: pramlintide, sibutramine, orlistat, zonisamide, topiramate, phentermine, naltrexone, bupropion, lorcaserin, metformin, or any GLP-1R agonists (either by prescription or as part of a clinical study).
* Prior exposure to maridebart cafraglutide or AMG 598 or currently receiving treatment in another investigational device or drug study, or less than 5 half-lives since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Female participants with a positive pregnancy test assessed at screening and/or day -2 by a serum pregnancy test and/or urine pregnancy test) or female participants who are breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 5 months after the last dose of maridebart cafraglutide.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use an acceptable method of contraception during treatment and for an additional 5 months after the last dose of maridebart cafraglutide.
* Male participants unwilling to abstain from donating sperm during treatment and for an additional 5 months after the last dose of maridebart cafraglutide.
* Participant has known sensitivity to maridebart cafraglutide or components thereof or a history of drug or other allergy that is in the opinion of the investigator or medical monitor (if appropriate), contraindicates their participation.
* Participant has a known sensitivity to GLP-1R agonists.
* Participant has known sensitivity to mammalian derived products.
* Participant has an allergy or known sensitivity to acetaminophen.
* Participant is unwilling or unable to limit alcohol consumption throughout the course of the study. Alcohol is prohibited 48 hours before day -2 and is limited to no more than to 2 drinks per day for males and 1 drink per day for females for the duration of the study (1 drink being equivalent to 12 ounces of regular beer, 8 to 9 ounces of malt liquor, 5 ounces of wine, or 1.5 ounces of 80 proof distilled spirits).
* Participant uses nicotine or tobacco containing products (including but not limited to: snuff, chewing tobacco, cigars, cigarettes, e-cigarettes, pipes, or nicotine patches) within 6 months before screening. Participant is unwilling or unable to abstain from nicotine or tobacco, cigars, cigarettes, pipes, or nicotine patches throughout the course of the study.
* Participant is tested positive for alcohol and/or drugs of abuse at screening.
* History of substance abuse (ie, alcohol, licit or illicit drugs) within 12 months before screening.
* Participant is unwilling to refrain from strenuous exercise (eg, heavy lifting, weight training, and aerobics) for 72 hours before each blood collection for clinical laboratory tests.
* Participant has donated or lost ≥ 500 mL of blood or plasma within 60 days of day -2.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.
* For participants in cohorts 7-10 and cohorts 12-13 only, the Patient Health Questionnaire-9 (PHQ-9) score of ≥ 10 up to day 1.
* For participants in cohorts 7-10 and 12-13 only, any suicidal ideation as identified by endorsement of (answered yes to) any of the items numbered 1-5 on the Columbia Suicide Severity Rating Scale (C-SSRS) up to day 1.
* For participants in cohorts 7-10 and 12-13 only, participant has systolic blood pressure ≥ 150 mm Hg or diastolic blood pressure ≥ 95 mm Hg on day 1. For each visit, if the initial blood pressure is elevated, the reading may be repeated once at least 15 minutes later and the lower of the 2 readings may be used.
* For participants in cohorts 7-10 and 12-13 only, a QTc of > 450 msec in males or > 470 msec in females up to day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, Anaheim, California
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, LLC, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Veniant MM, Lu SC, Atangan L, Komorowski R, Stanislaus S, Cheng Y, Wu B, Falsey JR, Hager T, Thomas VA, Ambhaikar M, Sharpsten L, Zhu Y, Kurra V, Jeswani R, Oberoi RK, Parnes JR, Honarpour N, Neutel J, Strande JL. A GIPR antagonist conjugated to GLP-1 analogues promotes weight loss with improved metabolic parameters in preclinical and phase 1 settings. Nat Metab. 2024 Feb;6(2):290-303. doi: 10.1038/s42255-023-00966-w. Epub 2024 Feb 5. PMID 38316982
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 110 participants were enrolled into this trial in the United States between August 2020 and November 2022.
Pre-assignment Details: This trial comprised three parts: Parts A and B were randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) phases, respectively; and part C was an open-label, modified, MAD phase.
Groups:
- Part A SAD Cohort 1 AMG 133: Participants received a single dose of 21 mg AMG 133 subcutaneously (SC).
- Part A SAD Cohort 2 AMG 133: Participants received a single dose of 70 mg AMG 133 SC.
- Part A SAD Cohort 3 AMG 133: Participants received a single dose of 140 mg AMG 133 SC.
- Part A SAD Cohort 4 AMG 133: Participants received a single dose of 280 mg AMG 133 SC.
- Part A SAD Cohort 5 AMG 133: Participants received a single dose of 560 mg AMG 133 SC.
- Part A SAD Cohort 6 AMG 133: Participants received a single dose of 70 mg AMG 133 intravenously (IV).
- Part A SAD SC Placebo (Cohorts 1-5, 11): Participants received a single dose of placebo SC.
- Part A SAD IV Placebo (Cohort 6): Participants received a single dose of placebo IV.
- Part B MAD Cohort 7 AMG 133: Participants received multiple doses of 140 mg AMG 133 SC every 4 weeks (Q4W).
- Part B MAD Cohort 8 AMG 133: Participants received multiple doses of 280 mg AMG 133 SC Q4W.
- Part B MAD Cohort 9 AMG 133: Participants received multiple doses of 560 mg AMG 133 SC Q4W.
- Part B MAD Cohort 10 AMG 133: Participants received multiple doses of 560 mg AMG 133 SC Q4W. This cohort included the use of digital health tools.
- Part B MAD Cohorts 7-9 Placebo: Participants received multiple doses of placebo SC Q4W.
- Part B MAD Cohort 10 Placebo: Participants received multiple doses of placebo SC Q4W. This cohort included the use of digital health tools.
- Part A SAD Cohort 11 AMG 133: Participants received a single dose of 840 mg AMG 133 SC.
- Part C MAD Cohort 12: Participants received 2 doses of 70 mg AMG 133 SC once weekly (QW), then 2 doses of 420 mg AMG 133 SC Q4W.
- Part C MAD Cohort 13: Participants received 4 doses of 70 mg AMG 133 SC QW, then 2 doses of 420 mg AMG 133 SC Q4W.
Period: Overall Study
Arm/Group | Part A SAD Cohort 1 AMG 133 | Part A SAD Cohort 2 AMG 133 | Part A SAD Cohort 3 AMG 133 | Part A SAD Cohort 4 AMG 133 | Part A SAD Cohort 5 AMG 133 | Part A SAD Cohort 6 AMG 133 | Part A SAD SC Placebo (Cohorts 1-5, 11) | Part A SAD IV Placebo (Cohort 6) | Part B MAD Cohort 7 AMG 133 | Part B MAD Cohort 8 AMG 133 | Part B MAD Cohort 9 AMG 133 | Part B MAD Cohort 10 AMG 133 | Part B MAD Cohorts 7-9 Placebo | Part B MAD Cohort 10 Placebo | Part A SAD Cohort 11 AMG 133 | Part C MAD Cohort 12 | Part C MAD Cohort 13
Started | 6 | 6 | 7 | 6 | 6 | 6 | 12 | 2 | 6 | 6 | 8 | 10 | 6 | 3 | 6 | 6 | 8
Completed | 6 | 5 | 5 | 6 | 5 | 5 | 11 | 2 | 5 | 5 | 3 | 5 | 5 | 3 | 5 | 6 | 4
Not Completed | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 5 | 5 | 1 | 0 | 1 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal of consent from study | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 3 | 0 | 0 | 1 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Part A SAD Cohort 1 AMG 133: Participants received a single dose of 21 mg AMG 133 SC.
- Part A SAD Cohort 6 AMG 133: Participants received a single dose of 70 mg AMG 133 IV.
- Part B MAD Cohort 7 AMG 133: Participants received multiple doses of 140 mg AMG 133 SC Q4W.
- Part C MAD Cohort 12: Participants received 2 doses of 70 mg AMG 133 SC QW, then 2 doses of 420 mg AMG 133 SC Q4W.
- Total: Total of all reporting groups
Arm/Group | Part A SAD Cohort 1 AMG 133 | Part A SAD Cohort 2 AMG 133 | Part A SAD Cohort 3 AMG 133 | Part A SAD Cohort 4 AMG 133 | Part A SAD Cohort 5 AMG 133 | Part A SAD Cohort 6 AMG 133 | Part A SAD SC Placebo (Cohorts 1-5, 11) | Part A SAD IV Placebo (Cohort 6) | Part B MAD Cohort 7 AMG 133 | Part B MAD Cohort 8 AMG 133 | Part B MAD Cohort 9 AMG 133 | Part B MAD Cohort 10 AMG 133 | Part B MAD Cohorts 7-9 Placebo | Part B MAD Cohort 10 Placebo | Part A SAD Cohort 11 AMG 133 | Part C MAD Cohort 12 | Part C MAD Cohort 13 | Total
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 12 | 2 | 6 | 6 | 8 | 10 | 6 | 3 | 6 | 6 | 8 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 7 | 6 | 6 | 6 | 12 | 2 | 6 | 6 | 8 | 10 | 6 | 3 | 6 | 6 | 8 | 109
  >=65 years | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 2 | 1 | 2 | 4 | 0 | 1 | 2 | 7 | 5 | 4 | 1 | 1 | 5 | 3 | 47
  Male | 1 | 5 | 4 | 4 | 5 | 4 | 8 | 2 | 5 | 4 | 1 | 5 | 2 | 2 | 5 | 1 | 5 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 0 | 0 | 5 | 2 | 2 | 4 | 4 | 10 | 2 | 3 | 5 | 1 | 2 | 45
  Not Hispanic or Latino | 5 | 4 | 6 | 5 | 6 | 6 | 7 | 0 | 4 | 2 | 4 | 0 | 4 | 0 | 1 | 5 | 6 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 5 | 3 | 0 | 5 | 4 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 2 | 33
  White | 4 | 4 | 2 | 3 | 5 | 1 | 8 | 2 | 2 | 5 | 7 | 10 | 5 | 3 | 5 | 2 | 4 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Part A: Maximum Observed Concentration (Cmax) of AMG 133
Description: The pharmacokinetic parameter estimates of intact and total AMG 133 after a single administration of AMG 133 were reported.
Time Frame: Cohort 1-5, 11: Day 1 predose and 1, 2, 4 and 8 hours postdose, Day 2, 3, 4, 5, 6, 7, 8, 15, 22, 29, 43, 57, 71, 92, 120 and 150. Cohort 6: Day 1 predose and 10 mins, 1, 2, 4 and 8 hours postdose, Day 2, 3, 4, 5, 6, 15, 22, 29, 43, 57, 71, 92, 120 and 150
Population: Pharmacokinetics analysis set: all participants who received at least 1 dose of AMG 133 for whom at least 1 pharmacokinetics parameter could be adequately estimated. Participants with data available at each timepoint are presented.
Measure: Geometric Mean (Standard Deviation); unit: µg/mL
Arm/Group | Part A SAD Cohort 1 AMG 133 | Part A SAD Cohort 2 AMG 133 | Part A SAD Cohort 3 AMG 133 | Part A SAD Cohort 4 AMG 133 | Part A SAD Cohort 5 AMG 133 | Part A SAD Cohort 6 AMG 133 | Part A SAD Cohort 11 AMG 133
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 4 | 6
µg/mL
  Intact AMG 133 | 1.31 (0.559) | 3.42 (1.18) | 6.09 (2.80) | 15.7 (11.4) | 35.8 (10.3) | 22.7 (4.10) | 41.5 (7.35)
  Total AMG 133 | 1.43 (0.614) | 3.68 (1.16) | 6.78 (3.16) | 17.1 (11.8) | 37.7 (12.5) | 22.9 (4.21) | 43.2 (7.07)

2. Secondary Outcome: Part B: Cmax of AMG 133
Description: The pharmacokinetic parameter estimates of intact and total AMG 133 after multiple administrations of AMG 133 were reported.
Time Frame: Cohorts 7-9: Day 1 (predose), Day 5, 7, 15, 22, 29 (predose), 36, 43, 50, 57 (predose), 61, 63, 71, 78, 85, 127, 169 and 207. Cohort 10: Day 1 (predose), Day 5, 7, 15, 22, 29 (predose), 36, 43, 50, 57 (predose), 63, 71, 78, 85, 169 and 207
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: µg/mL
Arm/Group | Part B MAD Cohort 7 AMG 133 | Part B MAD Cohort 8 AMG 133 | Part B MAD Cohort 9 AMG 133 | Part B MAD Cohort 10 AMG 133
Number analyzed (Participants) | 6 | 6 | 5 | 7
µg/mL
  Intact AMG 133 after dosing on Day 1: number analyzed (Participants) | 6 | 5 | 5 | 7
  Intact AMG 133 after dosing on Day 1 | 8.30 (2.59) | 14.5 (5.99) | 27.4 (12.4) | 17.8 (5.32)
  Total AMG 133 after dosing on Day 1: number analyzed (Participants) | 6 | 5 | 5 | 7
  Total AMG 133 after dosing on Day 1 | 8.75 (2.56) | 16.2 (6.52) | 30.1 (12.3) | 18.8 (5.15)
  Intact AMG 133 after dosing on Day 57: number analyzed (Participants) | 6 | 6 | 3 | 5
  Intact AMG 133 after dosing on Day 57 | 10.4 (2.19) | 21.9 (6.47) | 65.1 (20.4) | 27.2 (5.20)
  Total AMG 133 after dosing on Day 57: number analyzed (Participants) | 6 | 6 | 3 | 5
  Total AMG 133 after dosing on Day 57 | 13.1 (2.86) | 27.1 (8.12) | 80.8 (23.2) | 33.2 (6.77)

3. Secondary Outcome: Part A: Time of Maximum Observed Concentration (Tmax) of AMG 133
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Part A SAD Cohort 1 AMG 133 | Part A SAD Cohort 2 AMG 133 | Part A SAD Cohort 3 AMG 133 | Part A SAD Cohort 4 AMG 133 | Part A SAD Cohort 5 AMG 133 | Part A SAD Cohort 6 AMG 133 | Part A SAD Cohort 11 AMG 133
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 4 | 6
days
  Intact AMG 133 | 5.0 [2.9 to 6.9] | 4.9 [3.9 to 6.9] | 6.0 [5.0 to 13] | 5.8 [2.8 to 13] | 3.9 [2.9 to 6.9] | 0.025 [0.0049 to 0.044] | 5.4 [1.9 to 6.0]
  Total AMG 133 | 5.9 [4.0 to 6.9] | 4.9 [3.9 to 14] | 7.0 [6.0 to 13] | 6.9 [3.8 to 21] | 4.4 [2.9 to 6.9] | 0.043 [0.0049 to 0.044] | 5.9 [1.9 to 6.0]

4. Secondary Outcome: Part B: Tmax of AMG 133
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Part B MAD Cohort 7 AMG 133 | Part B MAD Cohort 8 AMG 133 | Part B MAD Cohort 9 AMG 133 | Part B MAD Cohort 10 AMG 133
Number analyzed (Participants) | 6 | 6 | 5 | 7
days
  Intact AMG 133 after dosing on Day 1: number analyzed (Participants) | 6 | 5 | 5 | 7
  Intact AMG 133 after dosing on Day 1 | 5.9 [3.8 to 6.2] | 6.0 [4.1 to 14] | 5.9 [3.9 to 15] | 4.0 [3.8 to 7.0]
  Total AMG 133 after dosing on Day 1: number analyzed (Participants) | 6 | 5 | 5 | 7
  Total AMG 133 after dosing on Day 1 | 6.0 [3.8 to 6.2] | 6.0 [4.1 to 14] | 5.9 [3.9 to 15] | 4.0 [3.8 to 14]
  Intact AMG 133 after dosing on Day 57: number analyzed (Participants) | 6 | 6 | 3 | 5
  Intact AMG 133 after dosing on Day 57 | 4.7 [4.1 to 15] | 4.3 [3.7 to 6.0] | 4.1 [4.0 to 5.1] | 6.0 [6.0 to 6.0]
  Total AMG 133 after dosing on Day 57: number analyzed (Participants) | 6 | 6 | 3 | 5
  Total AMG 133 after dosing on Day 57 | 5.6 [4.1 to 7.2] | 6.2 [3.7 to 14] | 4.1 [4.0 to 5.1] | 6.0 [6.0 to 6.0]

5. Secondary Outcome: Part A: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) of AMG 133
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Part A SAD Cohort 1 AMG 133 | Part A SAD Cohort 2 AMG 133 | Part A SAD Cohort 3 AMG 133 | Part A SAD Cohort 4 AMG 133 | Part A SAD Cohort 5 AMG 133 | Part A SAD Cohort 6 AMG 133 | Part A SAD Cohort 11 AMG 133
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 5 | 4 | 5
mcg*day/mL
  Intact AMG 133 | 39.0 (13.6) | 108 (35.2) | 230 (56.2) | 442 (263) | 762 (196) | 205 (67.9) | 1150 (280)
  Total AMG 133 | 56.4 (20.3) | 151 (51.2) | 300 (104) | 629 (375) | 1100 (321) | 264 (112) | 1720 (468)

6. Secondary Outcome: Part B: AUC From Day 0 to 28 (AUC0-28) of AMG 133
Description: The pharmacokinetic parameter estimates of intact and total AMG 133 after multiple administrations of AMG 133 were reported.
  This parameter shows the AUC over the 28-day dosing interval, both from Day 1 to Day 29 (predose) and from Day 57 to Day 85.
Time Frame: Cohorts 7-9: Day 1 (predose), Day 5, 7, 15, 22, 29 (predose), 57 (predose), 61, 63, 71, 78 and 85. Cohort 10: Day 1 (predose), Day 5, 7, 15, 22, 29 (predose), 57 (predose), 63, 71, 78 and 85
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Part B MAD Cohort 7 AMG 133 | Part B MAD Cohort 8 AMG 133 | Part B MAD Cohort 9 AMG 133 | Part B MAD Cohort 10 AMG 133
Number analyzed (Participants) | 6 | 5 | 4 | 5
mcg*day/mL
  Intact AMG 133 after dosing on Day 1 up to Day 29 | 149 (23.5) | 246 (95.5) | 594 (201) | 347 (28.7)
  Total AMG 133 after dosing on Day 1 up to Day 29: number analyzed (Participants) | 5 | 5 | 4 | 5
  Total AMG 133 after dosing on Day 1 up to Day 29 | 181 (26.0) | 300 (122) | 697 (244) | 419 (43.7)
  Intact AMG 133 after dosing on Day 57 up to Day 85: number analyzed (Participants) | 5 | 5 | 3 | 5
  Intact AMG 133 after dosing on Day 57 up to Day 85 | 214 (18.7) | 443 (136) | 1220 (432) | 512 (79.7)
  Total AMG 133 after dosing on Day 57 up to Day 85: number analyzed (Participants) | 5 | 5 | 3 | 5
  Total AMG 133 after dosing on Day 57 up to Day 85 | 297 (27.7) | 599 (224) | 1610 (624) | 691 (114)

7. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event (AE) which started on or after the first dose of AMG 133. Clinically significant changes in laboratory safety tests, vital signs and 12-lead electrocardiograms (ECGs) were included as AEs.
Time Frame: Part A: 150 days; Part B: 207 days; Part C Cohort 12: 193 days; Part C Cohort 13: 207 days
Population: Full analysis set: all randomized participants who received at least one dose of AMG 133 or placebo.
Measure: Number; unit: participants
Arm/Group | Part A SAD Cohort 1 AMG 133 | Part A SAD Cohort 2 AMG 133 | Part A SAD Cohort 3 AMG 133 | Part A SAD Cohort 4 AMG 133 | Part A SAD Cohort 5 AMG 133 | Part A SAD Cohort 6 AMG 133 | Part A SAD SC Placebo (Cohorts 1-5, 11) | Part A SAD IV Placebo (Cohort 6) | Part B MAD Cohort 7 AMG 133 | Part B MAD Cohort 8 AMG 133 | Part B MAD Cohort 9 AMG 133 | Part B MAD Cohort 10 AMG 133 | Part B MAD Cohorts 7-9 Placebo | Part B MAD Cohort 10 Placebo | Part A SAD Cohort 11 AMG 133 | Part C MAD Cohort 12 | Part C MAD Cohort 13
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 12 | 2 | 6 | 6 | 8 | 10 | 6 | 3 | 6 | 6 | 8
participants | 0 | 2 | 5 | 6 | 5 | 6 | 3 | 1 | 6 | 6 | 8 | 8 | 3 | 0 | 6 | 5 | 6

8. Secondary Outcome: Percentage of Participants With Anti-AMG 133 Antibody Formation
Description: The percentage of participants who developed anti-AMG 133 antibodies (binding and if positive, neutralizing to native GLP-1, when available) at any time was presented.
Time Frame: Part A Cohort 1-6 and 11: Up to Day 150. Part B Cohort 7-10 and Part C Cohort 13: Up to Day 207. Part C Cohort 12: Up to Day 193
Population: Full analysis set: all randomized participants who received at least one dose of AMG 133 or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Part A SAD Cohort 1 AMG 133 | Part A SAD Cohort 2 AMG 133 | Part A SAD Cohort 3 AMG 133 | Part A SAD Cohort 4 AMG 133 | Part A SAD Cohort 5 AMG 133 | Part A SAD Cohort 6 AMG 133 | Part B MAD Cohort 7 AMG 133 | Part B MAD Cohort 8 AMG 133 | Part B MAD Cohort 9 AMG 133 | Part B MAD Cohort 10 AMG 133 | Part A SAD Cohort 11 AMG 133 | Part C MAD Cohort 12 | Part C MAD Cohort 13
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 8 | 10 | 6 | 6 | 8
percentage of participants
  Binding antibody positive | 16.7 | 50.0 | 28.6 | 33.3 | 16.7 | 16.7 | 0.0 | 33.3 | 25.0 | 30.0 | 33.3 | 16.7 | 12.5
  Neutralizing antibody positive | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events, from enrollment to end of study; median duration (min, max) in months: 4.93 (0.13, 7.03). TEAEs from first dose of study drug until end of study; duration with median (min, max) in months: 4.93 (0.13, 7.03). TEAE time frame for Part A: 150 days; Part B: 207 days; Part C Cohort 12: 193 days; Part C Cohort 13: 207 days.
Description: Serious adverse events and other adverse events were reported for all participants who received at least one dose of study drug.
Arm/Group | Part A SAD Cohort 1 AMG 133 | Part A SAD Cohort 2 AMG 133 | Part A SAD Cohort 3 AMG 133 | Part A SAD Cohort 4 AMG 133 | Part A SAD Cohort 5 AMG 133 | Part A SAD Cohort 6 AMG 133 | Part A SAD SC Placebo (Cohorts 1-5, 11) | Part A SAD IV Placebo (Cohort 6) | Part B MAD Cohort 7 AMG 133 | Part B MAD Cohort 8 AMG 133 | Part B MAD Cohort 9 AMG 133 | Part B MAD Cohort 10 AMG 133 | Part B MAD Cohorts 7-9 Placebo | Part B MAD Cohort 10 Placebo | Part A SAD Cohort 11 AMG 133 | Part C MAD Cohort 12 | Part C MAD Cohort 13
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/12 | 0/2 | 0/6 | 0/6 | 0/8 | 0/10 | 0/6 | 0/3 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/12 | 0/2 | 0/6 | 0/6 | 0/8 | 0/10 | 0/6 | 0/3 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 5/7 | 6/6 | 5/6 | 6/6 | 3/12 | 1/2 | 6/6 | 6/6 | 8/8 | 8/10 | 3/6 | 0/3 | 6/6 | 5/6 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A SAD Cohort 1 AMG 133 (N=6) | Part A SAD Cohort 2 AMG 133 (N=6) | Part A SAD Cohort 3 AMG 133 (N=7) | Part A SAD Cohort 4 AMG 133 (N=6) | Part A SAD Cohort 5 AMG 133 (N=6) | Part A SAD Cohort 6 AMG 133 (N=6) | Part A SAD SC Placebo (Cohorts 1-5, 11) (N=12) | Part A SAD IV Placebo (Cohort 6) (N=2) | Part B MAD Cohort 7 AMG 133 (N=6) | Part B MAD Cohort 8 AMG 133 (N=6) | Part B MAD Cohort 9 AMG 133 (N=8) | Part B MAD Cohort 10 AMG 133 (N=10) | Part B MAD Cohorts 7-9 Placebo (N=6) | Part B MAD Cohort 10 Placebo (N=3) | Part A SAD Cohort 11 AMG 133 (N=6) | Part C MAD Cohort 12 (N=6) | Part C MAD Cohort 13 (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 4 | 4 | 5 | 6 | 3 | 0 | 5 | 4 | 8 | 3 | 1 | 0 | 5 | 4 | 6
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 5 | 5 | 2 | 0 | 0 | 4 | 5 | 6 | 7 | 0 | 0 | 4 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breath sounds absent (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 3 | 3 | 0 | 1 | 1 | 3
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT04478708/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT04478708/SAP_001.pdf